CLINICAL TRIAL: NCT05669560
Title: Efficacy of Hydrogen Peroxide Gel on Periodontal Ststus and Metabolic Control in Diabetic Patients: a Randomized Control Trial
Brief Title: Efficacy of Hydrogen Peroxide Gel on Periodontitis With Diabetes
Acronym: Peroxide gel
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The study team made the decision to not move forward with the study.
Sponsor: University of Oklahoma (Other)
Collaborators: Perio Protect LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Withdrawn
Record Dates: First submitted 2022-12-06; First posted 2023-01-03 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Periodontitis; Diabetes Mellitus
Keywords: non surgical periodontal therapy; scaling and root planing
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control group (No Intervention): Will receive SRP alone.
- Test group (Experimental): Will receive SRP + PerioProtect ™.
  Interventions: Combination Product: PerioProtect ™= plastic tray +1.7% hydrogen peroxide

INTERVENTIONS:
Combination Product: PerioProtect ™= plastic tray +1.7% hydrogen peroxide — Subjects will receive PerioProtect ™ in adjunct to mechanical therapy. 15minutes, twice a day, for 3 months.
  Arms: Test group

SUMMARY:
Periodontitis is a chronic infectious disease characterized by loss of tooth supporting periodontal structures and alveolar bone. In the U.S. and worldwide, periodontitis is the major cause of tooth loss in adults.

Type 2 Diabetes mellitus (T2DM) is a complex disease that affects 13-15 million Americans and is associated with a variety of serious complications. T2DM is well established as a strong systemic risk factor for periodontitis. The severity and prevalence of periodontitis is much higher in patients with diabetes. This relationship may be bi-directional.

DETAILED DESCRIPTION:
The primary treatment for periodontitis is scaling and root planing (SRP), which refers to the mechanical disruption and removal of bacteria and bacterial toxins from the affected tooth root surfaces. This procedure predictably reduces the bacterial load and produces marked improvement in clinical periodontal parameters, though not always complete resolution of the disease. Periodontal therapy may have some systemic benefits by reducing entry into the systemic circulation of pro inflammatory molecules and bacterial byproducts from the periodontal tissues. Since SRP alone is not always a completely effective treatment especially in advanced stages of periodontitis, a variety of adjunctive antimicrobial therapies such as local delivery of antimicrobial agents into periodontal pockets have been developed and employed to further reduce the bacterial load from periodontal pockets, with mixed results.

A recent innovation in the arena of local delivery antimicrobial agents is the PerioProtect ™ system (Perio Tray® and PerioGel® Perio Protect, St. Louis, MO). This consists of a closely fitting acrylic tray (similar to an athletic mouthguard), which is used to administer 1.7% hydrogen peroxide gel (Perio Gel®, QNT Anderson, Bismarck, ND) deep into the periodontal pocket and retain the gel in place for a sufficient time period (15 minutes) to effectively reduce the periodontal bacterial load. Studies to date have shown that when PerioProtect ™ is used as adjunct to conventional SRP, this system produces additional benefits in reducing the severity of periodontal disease. However, no studies have yet investigated the use of PerioProtect ™ in patients with T2DM and periodontitis.

Based on the concept of a bi-directional relationship of diabetes and periodontitis, the investigators hypothesize that successful management of periodontal infection in diabetics with the use of PerioProtect ™ will not only improve periodontal status, but also result in improved metabolic control of T2DM.

ELIGIBILITY:
Inclusion Criteria:

1. Adults >18 , <80 year old with moderate to severe periodontitis as defined by the Word workshop criteria having Type II diabetes mellitus with HbA1 C levels of >6.5%.
2. No SRP within the past 6 months.
3. Willingness to comply with study instructions and refrain from using oral hygiene products/ procedures outside the study.

Exclusion Criteria:

* The researcher believes that it is not in the patient's best interest to stay in the study
* Based on the exclusion criteria, the patient becomes ineligible to participate
* Patient's medical condition requires interventions which preclude involvement in the study
* Patient does not follow study related instructions
* The study is suspended or canceled

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-20 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of HbA1C measured in percentage. | Measured at baseline
  To investigate the efficacy of locally delivered 1.7% hydrogen peroxide gel (Perio Gel®)as an adjunct to mechanical periodontal therapy on glycemic control in periodontitis patients with Type 2 diabetes mellitus.
Change of HbA1C measured in percentage. | Measured at 3 months
  To investigate the efficacy of locally delivered 1.7% hydrogen peroxide gel (Perio Gel®)as an adjunct to mechanical periodontal therapy on glycemic control in periodontitis patients with Type 2 diabetes mellitus.
Change of HbA1C measured in percentage. | Measured at 6 months
  To investigate the efficacy of locally delivered 1.7% hydrogen peroxide gel (Perio Gel®)as an adjunct to mechanical periodontal therapy on glycemic control in periodontitis patients with Type 2 diabetes mellitus.
Change of HbA1C measured in percentage. | Measured at 9 months
  To investigate the efficacy of locally delivered 1.7% hydrogen peroxide gel (Perio Gel®)as an adjunct to mechanical periodontal therapy on glycemic control in periodontitis patients with Type 2 diabetes mellitus.

SECONDARY OUTCOMES:
Change in Probing Pocket Depth(mm) | Measured at baseline, 3, 6, 9months.
  To determine if the use of PerioProtect ™ as an adjunct to mechanical therapy produces additional improvement in periodontal status as compared to conventional periodontal therapy (SRP) alone.
Change in Bleeding On Probing(%) | Measured at baseline, 3, 6, 9months.
  To determine if the use of PerioProtect ™ as an adjunct to mechanical therapy produces additional improvement in periodontal status as compared to conventional periodontal therapy (SRP) alone.
Change in Plaque Index (0-3). | Measured at baseline, 3, 6, 9months.
  To determine if the use of PerioProtect ™ as an adjunct to mechanical therapy produces additional improvement in periodontal status as compared to conventional periodontal therapy (SRP) alone.
Change in Clinical attachment levels(mm). | Measured at baseline, 3, 6, 9months.
  To determine if the use of PerioProtect ™ as an adjunct to mechanical therapy produces additional improvement in periodontal status as compared to conventional periodontal therapy (SRP) alone.

CONTACTS AND LOCATIONS:
Overall Officials: John Dmytryk, DDS, PhD, Study Chair — The University of Oklahoma, College of Dentistry, Division in Periodontics

IPD SHARING:
Plan to Share IPD: Undecided